CLINICAL TRIAL: NCT00900367
Title: Nutrition Modulated Metabolism as a Disease Risk Factor
Brief Title: Nutrition-Related Biomarkers in Predicting Breast Cancer Risk in Women
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bruce Kristal, Associate Professor, Brigham and Women's Hospital
Other Study IDs: CDR0000583255; BWH-BRC322; R01CA102536 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Chromatography, High Pressure Liquid; Spectrum Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — we have only plasma, NHS has DNA samples.
  Study is nested case control, so retrospective with respect to individual inclusion, prospective with respect to sample collected before disease. Enrollment is approximate as it includes samples that will be drpped, eg for QC resons
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: high performance liquid chromatography
Other: laboratory biomarker analysis
Procedure: spectroscopy

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about nutrition-related changes that identify biomarkers related to cancer. It may also help doctors predict a woman's risk of developing breast cancer.

PURPOSE: This laboratory study is looking at nutrition-related biomarkers in predicting breast cancer risk in women.

DETAILED DESCRIPTION:
OBJECTIVES:

* To complete characterization of metabolic serotypes based on the metabolome, and to adapt these profiles for human epidemiological studies.
* To determine the extent to which metabolic profiles that are reflective of or independent of long-term caloric intake predict breast cancer risk in nested case-control studies.
* To identify critical serum metabolites.

OUTLINE: Laboratory studies, including metabolome profiling by high performance liquid chromatography; and small molecule identification by mass spectroscopy, are performed on previously collected blood samples.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Confirmed breast cancer that was diagnosed at least 2 years after blood sample collection (case)

    * No prior diagnosis of cancer
  * Healthy participant (control)
* Enrolled in the Nurses' Health Study
* Banked blood samples available
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women enrolled in the NHS I study; Group selected by Drs. Willett and Hankinson
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2005-07; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Generation of metabolome profiles that reflect nutritional status | ongoing
Utility of rat metabolome profiles for human epidemiological studies | ongoing
Utility of metabolome profiles in predicting relative risk of developing breast cancer | ongoing
Identification of critical serum metabolites | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Bruce S. Kristal, PhD, Study Chair — Brigham and Women's Hospital
Locations (1):
- Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts, United States